CLINICAL TRIAL: NCT05969587
Title: Compare the Efficacy and Safety Profile of Cysteamine and Hydroquinone in Melasma as Topical Application
Brief Title: Cysteamine Compared to Hydroquinone in Melasma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH108-REC1-145
Record Dates: First submitted 2023-07-05; First posted 2023-08-01 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients treated with 5% cysteamine cream (Experimental)
  Interventions: Combination Product: 5% cysteamine cream
- patients treated with a combination of 4% hydroquinone cream and 0.06% betamethasone valerate (Active Comparator)
  Interventions: Combination Product: hydroquinone cream group

INTERVENTIONS:
Combination Product: 5% cysteamine cream — 5% cysteamine cream (Cyspera®) was acquired from Scientis APAC Pte. Ltd. (Singapore, Singapore).Subjects were instructed to thinly apply the designated creams to their whole face every evening 15 minutes after cleansing their faces with a designated soap and the application of a skin moisturizer. The cysteamine cream was washed off 15 minutes after application
  Arms: patients treated with 5% cysteamine cream
Combination Product: hydroquinone cream group — 4% w/w hydroquinone cream (Melquine™) and 0.06% w/w betamethasone valerate cream (Rinderon®-V; equivalent to 0.05% betamethasone) were acquired from Sinphar Pharmaceutical Co., Ltd. (Yilan, Taiwan). Subjects were instructed to thinly apply the designated creams to their whole face every evening 15 minutes after cleansing their faces with a designated soap and the application of a skin moisturizer. Subjects in the hydroquinone cream group were told to apply a 2:1 ratio of the hydroquinone and betamethasone creams. The hydroquinone/betamethasone creams were left on the skin until the following morning.
  Arms: patients treated with a combination of 4% hydroquinone cream and 0.06% betamethasone valerate

SUMMARY:
Melasma is an acquired pigmentary disorder of symmetrical hyperpigmentation appearing as variable darkness macules and patches over the forehead, cheeks, and chin, even sun-exposed areas of the body. Melasma is predominantly affects women but men can also be affected. Melasma is commonly seen in Asia, where patients with Fitzpatrick skin types III and IV, and areas of high ultraviolet radiation. It is challenging and difficult to treat melasma for its refractory and recurrent nature. There is a variety of therapeutic approaches include topical medication with Kligman's formula, oral medication, chemical peels, lasers, and light therapy.

Cysteamine (b-mercaptoethylamine) hydrochloride is the stable amino-thiol that acts as an antioxidant. It can be naturally produced in the human body and is a degrada-tion product of the amino acid L-cysteine. It has been known to be a potent depigmenting agent for about five decades. The mechanism of cysteamine for depimentation is not through melanotoxicity, which is the major depigmentation mechanism of hydro-quinone. Exogenous ochronsis is the major concern about the long-term use of hydro-quinone. Cysteamine is a thiolic compound that inhibit tyrosinase and peroxidase activity of melanocytes and produce notably greater amounts of pheomelanin but less eumelanin. In addition, thiols can act as a chelating agent of iron and copper ions Fenton reaction during pigment synthesis. Thols can also scavenge dopaquinone and deplete dopaquinone from the melanogenesis pathway. Then, higher levels of intra-cellular glutathione augmented by cysteamine cause the melanogenesis to proceed at a slower rate by shifting eumelanogenesis to pheomelanin synthesis.

Since new technology permits reduction of the sulfur-odour of cysteamine hydro-chloride, cysteamine 5% cream permit the use in topical depigmenting preparations. Considerable efficacy and safety of cysteamine 5% cream in the treatment of epidermal melasma were confirmed by comprehensive measurements in previous well-controlled studies.

However, the depigmenting efficacy of cysteamine compared with hydroquinone has never been evaluated. In addition, durability of the depigmenting efficacy has never been reported and the maintenance usage the cysteamine 5% cream has never yet been studied. In the present study, the investigators evaluate the efficacy of cysteamine 5% cream with hy-droquinone 4% cream in treating melasma and provide the maintenance regimen of cys-teamine 5% cream for Asian patients with melasma.

ELIGIBILITY:
Inclusion Criteria:

* a history of epidermal type melasma as diagnosed by a board-certified dermatologist
* above the age of 20 years
* Fitzpatrick skin type II-V

Exclusion Criteria:

* pregnant
* breastfeeding
* currently receiving oral contraceptive pill or hormonal therapy
* have received topical hydroquinone, retinoid, tranexamic acid, or steroid treatment within the past month
* have received laser therapy or any other phototherapy within the past three months
* a history of allergic reactions to hydroquinone or cysteamine
* other pigmentary disorders of the face
* systemic diseases that may affect pigmentation of the face (such as systemic lupus erythematosus, jaundice, end-stage renal disease)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Change of Baseline Melasma Area and Severity Index (MASI) scores | Measurements were done at baseline and during subsequent follow-ups at 4 weeks and 12 weeks.
  MASI scores were computed according to the formula proposed by Kimbrough-Green et al. (1994) , whereby the surface area is graded as 0 (no involvement), 1 (< 10% involvement), 2 (10-29% involvement), 3 (30-49% involvement), 4 (50-69% involvement), 5 (70-89% involvement), and 6 (90-100% involvement). Darkness and homogeneity were graded as 0 (absent), 1 (slight), 2 (mild), 3 (marked), and 4 (severe).

SECONDARY OUTCOMES:
Erythema, melanin content, and luminance | Measurements were done at baseline and during subsequent follow-ups at 4 weeks and 12 weeks.
  Erythema, melanin content, and luminance at three predesignated regions of the face were measured with the skin color probe of DermaLab® Combo (Cortex Technology, Hadsund, Denmark), utilizing two high intensity white LED light sources and four 16-color sensor elements. Erythema and melanin content were measured in arbitrary units between 0 and 99.9, while luminance was derived from the CIELAB color space values whereby the lightness value is calculated from a 100% relative luminance of white and an offset near black. VISIA® Skin Analysis System (Canfield Scientific, Fairfield, New Jersey) was then used to take frontal and lateral cross-polarized photographs of the bilateral face in both the visible light and ultraviolet spectrum at fixed angles, distances, and camera settings. The measurement units used above are all arbitrary units.
Spots, wrinkles, skin texture, pore numbers, UV spots, brown spots, red areas, and porphyrins | Measurements were done at baseline and during subsequent follow-ups at 4 weeks and 12 weeks.
  The standardized photographs were then evaluated for spots, wrinkles, skin texture, pore numbers, UV spots, brown spots, red areas, and porphyrins by comparing them to Canfield's worldwide skin feature database and calculating the percentile ranking for each feature, whereby a higher percentile score indicates better skin condition.
patient satisfaction on depigmentation and overall satisfaction | The satisfaction scale was evaluated after 12 week of treatment.
  During follow-up, patient satisfaction on depigmentation and overall satisfaction were evaluated and scored on a scale between one to five, with one being extremely dissatisfied and five being extremely satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan